CLINICAL TRIAL: NCT03792659
Title: Exploring Outcomes and Characteristics of Myasthenia Gravis: The EXPLORE MG Registry
Brief Title: The EXPLORE MG Registry for Myasthenia Gravis
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1602017284
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples Without DNA — 100 cc (less than 1/2 cup) of blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurological Outpatients: Participants in this group will be recruited from the outpatient clinical population at the Yale University Department of Neurology. Treating physicians will make the initial determination of patients' potential eligibility to participate in the study.
  Interventions: Other: Blood Sample Draw

INTERVENTIONS:
Other: Blood Sample Draw — Approximately 100 cc (less than 1/2 cup) of blood will be drawn from both groups.

SUMMARY:
The purpose of this study is to create a Yale University Department of Neurology Myasthenia Gravis (MG) registry that will be used for current and future research projects involving the study of Myasthenia Gravis.

DETAILED DESCRIPTION:
This registry will allow for the research of several mechanisms of Myasthenia Gravis (MG) by studying peripheral blood, stool, disease status and course, and treatment of subjects with MG. The EXPLORE-MG Registry focuses on varied aspects of MG such as disease management, health care utilization, health costs, disease characteristics, and diagnostic tools. As such, it will aid in a broader understanding of MG, while providing a registry from which questions about the disease may be better answered.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with Myasthenia Gravis presenting to the Yale Department of Neurology for clinical care or research interventions will be invited to donate their biological specimens/clinical data.

Exclusion Criteria:

* Failure to meet the Inclusion Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be 18 years of age or older with a clinical diagnosis of a Myasthenia Gravis.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-03-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
The number of successful blood draws will be reported at the conclusion of the sample collection | 8 years
  Successful Collection of Blood

SECONDARY OUTCOMES:
The number of stool samples collected will be reported at the conclusion of the sample | 8 years
  Count of Stool Samples

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nowak, MD, MS, Principal Investigator — Assistant Professor, Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anil R, Kumar A, Alaparthi S, Sharma A, Nye JL, Roy B, O'Connor KC, Nowak RJ. Exploring outcomes and characteristics of myasthenia gravis: Rationale, aims and design of registry - The EXPLORE-MG registry. J Neurol Sci. 2020 Jul 15;414:116830. doi: 10.1016/j.jns.2020.116830. Epub 2020 Apr 16. PMID 32388060